CLINICAL TRIAL: NCT03173677
Title: Monocyte Differentiation and Macrophage Polarization in Circulation in Response to Macronutrient Intake in Healthy Humans: A Randomized Clinical Study
Brief Title: Macrophage Polarization in Response to Macronutrient Intake in Healthy Humans: A Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud Bin Abdulaziz University for Health Sciences (Other)
Responsible Party: Principal Investigator, Ahmad Aljada, Professor of Biochemistry, King Saud Bin Abdulaziz University for Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SP15/026
Record Dates: First submitted 2017-05-28; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Atherosclerosis
Keywords: Mononuclear cells; Whey proteins; Metabolically-Activated Macrophage; Macrophage Polarization; Macronutrients
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lipid intake (Active Comparator): 12 subjects had 300 Calories of lipids or 300 mL of water. Blood samples were drawn at 0, 1, 2, and 3 hrs post intake. There was a one week period between the 2 intakes.
  Interventions: Dietary Supplement: Lipid Intake
- Glucose intake (Active Comparator): 12 subjects had 300 Calories of glucose or 300 mL of water. Blood samples were drawn at 0, 1, 2, and 3 hrs post intake. There was a one week period between the 2 intakes.
  Interventions: Dietary Supplement: Glucose intake
- Protein intake (Active Comparator): 12 subjects had 300 Calories Whey protein intake or 300 mL of water. Blood samples were drawn at 0, 1, 2, and 3 hrs post intake. There was a one week period between the 2 intakes.
  Interventions: Dietary Supplement: Protein intake

INTERVENTIONS:
Dietary Supplement: Lipid Intake — 90 grams whipping cream, 31.5 grams fat, 1.7 grams protein, and 2.25 grams carbohydrate
  Arms: Lipid intake
Dietary Supplement: Glucose intake — 300 calories of glucose
  Arms: Glucose intake
Dietary Supplement: Protein intake — Isopure unflavored Whey proteins isolate (WPI) powder containing 26 grams per serving of 100% WPI, stripped of fat, carbs, fillers, sugars, and lactose
  Arms: Protein intake

SUMMARY:
Macrophages can exhibit distinct phenotypes and functions in response to stimuli and can polarize into one of three distinct phenotypes: a pro-inflammatory (M1), an anti-inflammatory pro-tissue (M2) and metabolically-activated (MMe) macrophage phenotypes. Thirty-six healthy volunteers were recruited and randomized into one of three macronutrient intake groups (glucose, lipids, proteins). This study measured the effects of macronutrient intake on the macrophage differentiation.

DETAILED DESCRIPTION:
Thirty-six normal healthy adult volunteers of normal weight were recruited into the study. All were normotensive, had a normal lipid profile, normal renal and liver function tests, and were not on any medications. All subjects gave their written, informed consent. Institutional Review Board (IRB) of the Ministry of National Guard Health Affairs (MNGHA) approved the study protocol. The 36 participants were randomly assigned by the primary investigator (PI) following simple randomization procedure (computerized random numbers) to three different groups, each received one type of macronutrient (Glucose, whey proteins or lipids). Following an overnight fast, a baseline blood sample was taken. Subjects were then given either 300 calories of glucose (NERL Trutol 75) or lipids (90 grams whipping cream, 31.5 grams fat, 1.7 grams protein and 2.25 grams carbohydrate) or protein (Isopure unflavored Whey proteins isolate (WPI) powder containing 26 grams per serving of 100% WPI, stripped of fat, carbs, fillers, sugars and lactose) solution over 5 minutes. Cream and protein preparations were diluted with water up to 300 mL solutions. Further blood samples were obtained at 1, 2 and 3 hours after the macronutrient intake. Subjects, either one week before or after the macronutrient challenge, were given 300 mL of water to drink in the fasting state. Blood samples were obtained before and at 1, 2 and 3 h after water intake as well. Each subject served as his/her own control and was randomly given macronutrient or water intake.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (BMI 18.5-25)
* Healthy adults evident by: physical examination, normal lipid profile, normal renal and liver function tests.

Exclusion Criteria:

* Renal disease
* Hepatic disease
* Cardiovascular disease
* Using multivitamins
* Using NSAIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-04-24 (Actual); Study Completion 2016-04-29 (Actual)

PRIMARY OUTCOMES:
Detection of markers of M1 and M2 macrophages | Subject recruitment, enrollment and sample collection were carried out in a period of 3 months. Baseline blood samples were drawn before the caloric or water intake, and subsequent blood samples were drawn at 1-, 2- and 3-hour intervals post the intake
  The following markers were used to detect M1 and M2 macrophages (M1:CD86, IL-6, CD11c, and CD169, and M2: CD206, CD163, and CD36)

CONTACTS AND LOCATIONS:
Overall Officials: Awad Alshahrani, MD, Principal Investigator — Ministry of Natioanl Guard Health Affairs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Italiani P, Boraschi D. From Monocytes to M1/M2 Macrophages: Phenotypical vs. Functional Differentiation. Front Immunol. 2014 Oct 17;5:514. doi: 10.3389/fimmu.2014.00514. eCollection 2014. PMID 25368618
- [Background] Martinez FO, Gordon S. The M1 and M2 paradigm of macrophage activation: time for reassessment. F1000Prime Rep. 2014 Mar 3;6:13. doi: 10.12703/P6-13. eCollection 2014. PMID 24669294
- [Background] Billiau A, Matthys P. Interferon-gamma: a historical perspective. Cytokine Growth Factor Rev. 2009 Apr;20(2):97-113. doi: 10.1016/j.cytogfr.2009.02.004. Epub 2009 Mar 5. PMID 19268625
- [Background] Guha M, Mackman N. LPS induction of gene expression in human monocytes. Cell Signal. 2001 Feb;13(2):85-94. doi: 10.1016/s0898-6568(00)00149-2. PMID 11257452
- [Background] Feghali CA, Wright TM. Cytokines in acute and chronic inflammation. Front Biosci. 1997 Jan 1;2:d12-26. doi: 10.2741/a171. PMID 9159205
- [Background] Stein M, Keshav S, Harris N, Gordon S. Interleukin 4 potently enhances murine macrophage mannose receptor activity: a marker of alternative immunologic macrophage activation. J Exp Med. 1992 Jul 1;176(1):287-92. doi: 10.1084/jem.176.1.287. PMID 1613462
- [Background] Hotamisligil GS, Shargill NS, Spiegelman BM. Adipose expression of tumor necrosis factor-alpha: direct role in obesity-linked insulin resistance. Science. 1993 Jan 1;259(5091):87-91. doi: 10.1126/science.7678183.
- [Background] Visser M, Bouter LM, McQuillan GM, Wener MH, Harris TB. Elevated C-reactive protein levels in overweight and obese adults. JAMA. 1999 Dec 8;282(22):2131-5. doi: 10.1001/jama.282.22.2131. PMID 10591334
- [Background] Fried SK, Bunkin DA, Greenberg AS. Omental and subcutaneous adipose tissues of obese subjects release interleukin-6: depot difference and regulation by glucocorticoid. J Clin Endocrinol Metab. 1998 Mar;83(3):847-50. doi: 10.1210/jcem.83.3.4660. PMID 9506738
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Stoger JL, Gijbels MJ, van der Velden S, Manca M, van der Loos CM, Biessen EA, Daemen MJ, Lutgens E, de Winther MP. Distribution of macrophage polarization markers in human atherosclerosis. Atherosclerosis. 2012 Dec;225(2):461-8. doi: 10.1016/j.atherosclerosis.2012.09.013. Epub 2012 Sep 26. PMID 23078881
- [Background] Mohanty P, Ghanim H, Hamouda W, Aljada A, Garg R, Dandona P. Both lipid and protein intakes stimulate increased generation of reactive oxygen species by polymorphonuclear leukocytes and mononuclear cells. Am J Clin Nutr. 2002 Apr;75(4):767-72. doi: 10.1093/ajcn/75.4.767. PMID 11916766